CLINICAL TRIAL: NCT03285607
Title: Phase I Study of MCS110 Combined With Neoadjuvant Dose-Dense Doxorubicin, Cyclophosphamide, and Weekly Paclitaxel in Patients With Hormone-Receptor Positive and HER2- Breast Cancer
Brief Title: MCS110 Combined With Neoadjuvant Doxorubicin, Cyclophosphamide, and Weekly Paclitaxel in Patients With Hormone-Receptor Positive and HER2- Breast Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Drug provider decided not to move forward with the study.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201711073; MCS110ZUS02T (Other: Novartis Pharmaceuticals)
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer; Cancer of Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Doxorubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Level 1:MCS110/Doxorubicin/Cyclophosphamide/Paclitaxel (Experimental): * MCS110 will be administered intravenously over 60 minutes (up to 120 minutes permitted) on a 28-day cycle. The dose of MCS110 given will depend on the dose level to which a given patient is enrolled.
  * The standard neoadjuvant chemotherapy regimen of dose-dense doxorubicin/ cyclophosphamide followed by weekly paclitaxel consists of:
    * doxorubicin 60 mg/m^2 IV Q2W during Weeks 1 through 8 (total of 4 doses)
    * cyclophosphamide 600 mg/m^2 Q2W during Weeks 1 through 8 (total of 4 doses)
    * paclitaxel 80 mg/m^2 IV QW during Weeks 9 through 20 (total of 12 doses)
  * Surgery will be performed approximately 4-6 weeks after the end of the last cycle of treatment (Week 20-22). It is outside the scope of this study as part of each patient's standard of care. Both types of surgery (lumpectomy or mastectomy) are allowed. The decision on surgical approach and timing will be at the discretion of the treating surgeon.
  Interventions: Biological: MCS110; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Procedure: Bone marrow aspirate; Procedure: Peripheral blood samples; Procedure: Tumor tissue
- Dose Level 2:MCS110/Doxorubicin/Cyclophosphamide/Paclitaxel (Experimental): * MCS110 will be administered intravenously over 60 minutes (up to 120 minutes permitted) on a 28-day cycle. The dose of MCS110 given will depend on the dose level to which a given patient is enrolled.
  * The standard neoadjuvant chemotherapy regimen of dose-dense doxorubicin/ cyclophosphamide followed by weekly paclitaxel consists of:
    * doxorubicin 60 mg/m^2 IV Q2W during Weeks 1 through 8 (total of 4 doses)
    * cyclophosphamide 600 mg/m^2 Q2W during Weeks 1 through 8 (total of 4 doses)
    * paclitaxel 80 mg/m^2 IV QW during Weeks 9 through 20 (total of 12 doses)
  * Surgery will be performed approximately 4-6 weeks after the end of the last cycle of treatment (Week 20-22). It is outside the scope of this study as part of each patient's standard of care. Both types of surgery (lumpectomy or mastectomy) are allowed. The decision on surgical approach and timing will be at the discretion of the treating surgeon.
  Interventions: Biological: MCS110; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Procedure: Bone marrow aspirate; Procedure: Peripheral blood samples; Procedure: Tumor tissue
- Dose Expansion:MCS110/Doxorubicin/Cyclophosphamide/Paclitaxel (Experimental): * MCS110 will be administered intravenously over 60 minutes (up to 120 minutes permitted) on a 28-day cycle. The dose of MCS110 given will depend on the dose level to which a given patient is enrolled.
  * The standard neoadjuvant chemotherapy regimen of dose-dense doxorubicin/ cyclophosphamide followed by weekly paclitaxel consists of:
    * doxorubicin 60 mg/m^2 IV Q2W during Weeks 1 through 8 (total of 4 doses)
    * cyclophosphamide 600 mg/m^2 Q2W during Weeks 1 through 8 (total of 4 doses)
    * paclitaxel 80 mg/m^2 IV QW during Weeks 9 through 20 (total of 12 doses)
  * Surgery will be performed approximately 4-6 weeks after the end of the last cycle of treatment (Week 20-22). It is outside the scope of this study as part of each patient's standard of care. Both types of surgery (lumpectomy or mastectomy) are allowed. The decision on surgical approach and timing will be at the discretion of the treating surgeon.
  Interventions: Biological: MCS110; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel; Procedure: Bone marrow aspirate; Procedure: Peripheral blood samples; Procedure: Tumor tissue

INTERVENTIONS:
Biological: MCS110 — -MCS110 is an IgG1/κ humanized monoclonal antibody directed against human macrophage colony stimulating factor
Drug: Doxorubicin — -Standard of care
  Other Names: Adriamycin®
Drug: Cyclophosphamide — -Standard of care
  Other Names: Cytoxan; CPM; CTX; CYT
Drug: Paclitaxel — -Standard of care
  Other Names: Taxol
Procedure: Bone marrow aspirate — -Time of enrollment and at time of surgery
Procedure: Peripheral blood samples — -Time of enrollment and at time of surgery
Procedure: Tumor tissue — -Time of enrollment and at time of surgery

SUMMARY:
In patients with locally advanced hormone receptor positive (HR+)/HER2- breast cancer, neoadjuvant chemotherapy produces a pathologic complete response rate (pCR) of only 9-15%, and late recurrences often occur despite neoadjuvant chemotherapy. Therefore, there is an unmet clinical need to improve the outcomes of these patients. Tumor-associated macrophages (TAM) infiltration leads to poor outcomes in breast cancer patients by promoting angiogenesis, activating epithelial-mesenchymal transition, degrading the extracellular matrix, and suppressing the anti-tumor immune response. Pre-clinical studies, as summarized above, have shown that the breast cancer immune microenvironment may be reprogrammed by targeting colony-stimulating factor-1 (CSF-1) to decrease TAM infiltration and increase CD8+ TIL infiltration, in order to foster antitumor immunity and improve response to therapy.

Here, the investigators propose a phase I dose-escalation study in patients with locally advanced HR+/HER2- breast cancer to determine the feasibility of adding MCS110, a CSF-1 inhibitor, to the standard neoadjuvant chemotherapy regimen of dose-dense doxorubicin, cyclophosphamide followed by paclitaxel. The investigators will also include a dose expansion cohort for preliminary efficacy analysis and correlative studies. The investigators propose that if they can decrease the TAM-induced immunosuppression and TAM-induced chemoresistance observed in breast cancer patients, then the patients' own immune system could find and destroy the dormant and resistant tumor cells, and combined with enhanced chemotherapy efficacy, the investigators will see durable remissions and long term cures.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed ER+ HER2- breast cancer. ER-positivity is to follow local guidelines. If IHC HER2 is 2+, a negative FISH test is required.
* Clinical stage II or stage III (by AJCC 7th edition) breast cancer eligible for neoadjuvant chemotherapy with complete surgical excision of the breast cancer after neoadjuvant therapy as the treatment goal.
* Clinically positive axillary lymph nodes.
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 x institutional upper limit of normal (IULN)
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Creatinine ≤ 1.5 x IULN
  * PT/INR ≤ 1.5 x IULN (for participants on anticoagulation therapy, ≤ 1.5 x baseline value)
  * aPTT ≤ 1.5 x IULN (for participants on anticoagulation therapy, ≤ 1.5 x baseline value)
* Adequate cardiac function as defined below:

  * LVEF ≥ 50%
  * QTC ≤ 470 msec for females and ≤ 450 msec for males
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry, for the duration of study participation, and for 90 days after the last dose of MCS110. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 4 month after completion of MCS110 administration.
* Ability to understand and willingness to sign an Institutional Review Board (IRB) approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Presence of metastatic disease.
* Therapy for underlying malignancy within 2 weeks prior to start of study treatment.
* A history of other malignancy ≤ 3 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Bilateral or inflammatory breast cancer.
* Currently receiving any other investigational agents.
* Receiving immunosuppressive agents or > 10 mg daily prednisone or equivalent of corticosteroids.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to MCS110, doxorubicin, cyclophosphamide, paclitaxel, or other agents used in the study.
* Known hypersensitivity to monoclonal antibodies.
* Personal or family history of long QT syndrome.
* Evidence of retinal pathology on ophthalmologic examination that is considered a risk factor for neurosensory retinal detachment / central serous chorioretinopathy (CSCR), retinal vein occlusion (RVO), or neovascular macular degeneration.
* Diagnosis of any type of muscle disease that may result in CK elevation.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia. Clinically significant cardiovascular disease within 6 months of screening.
* Presence of any Common Terminology Criteria for Adverse Events (CTCAE) grade 2 or greater toxicity.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.
* Known history of human immunodeficiency virus or infection with hepatitis requiring antiviral therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-30 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of regimen | Completion of cycle 1 (28 days) for all patients
  * The maximum tolerated dose (MTD) is defined as the dose level at which <1 patients of a cohort (of 3 to 6 patients) experience dose-limiting toxicity during the first cycle.
  * A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value of CTCAE Grade ≥ 3 assessed as unrelated to disease, disease progression, intercurrent illness, or concomitant medications that occurs within the first cycle of treatment with the combination treatment and meets any of the criteria outlined.

SECONDARY OUTCOMES:
Safety and tolerability of regimen as measured by grade and number of adverse events experienced per participant | 30 days after completion of treatment (approximately 24 weeks)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Pathologic complete response-rate (pCR) | At the time of surgery (approximately 20 weeks)
  -Pathologic complete response (pCR) is defined as no histology evidence of invasive tumor cells in the surgical breast specimen and sentinel or axillary lymph nodes. All eligible patients who have completed neoadjuvant therapy and have subsequently undergone surgery are included in the analysis of pCR.
Residual invasive tumor size (RITS) | At the time of surgery (approximately 20 weeks)
  -Residual invasive tumor size (RITS) is histopathologically assessed by the largest dimension of the dominant invasive tumor focus from the surgical specimen. In cases in which there was no residual invasive tumor, the RITS will be 0 mm. In cases in which multifocal pathology is present, the largest dimension of the residual invasive tumor focus will be recorded.
Number of positive axillary lymph nodes | At the time of surgery (approximately 20 weeks)
  -Number of positive axillary lymph nodes is defined as number of resected lymph nodes with axillary nodal micrometastases (>0.2-<2 mm) or overt metastases (⩾2 mm).

CONTACTS AND LOCATIONS:
Overall Officials: Leonel Hernandez-Aya, M.D., Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu